CLINICAL TRIAL: NCT06340412
Title: Effects of Intact and Disrupted Milk Fat Globule Membrane on Postprandial Metabolic Response to High-fat Dairy in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MFGM-FOR-HEALTH
Record Dates: First submitted 2024-03-06; First posted 2024-04-01 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-02

CONDITIONS: Postprandial Lipid Metabolism
Keywords: Milk fat globule membrane
MeSH Terms: interventions — Breakfast; Lunch

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded, controlled, crossover trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-fat meal with intact MFGM (Experimental)
  Interventions: Dietary Supplement: Sandwich with butter-like dairy product (40g milk fat) with intact MFGM. One sandwich for breakfast and one sandwich for lunch.
- High-fat meal with destroyed MFGM (Experimental)
  Interventions: Dietary Supplement: Sandwich with butter-like dairy product (40g milk fat) with disrupted MFGM. One sandwich for breakfast and one sandwich for lunch.
- High-fat meal without MFGM (Experimental)
  Interventions: Dietary Supplement: Sandwich with butter-like dairy product (40g milk fat) without MFGM. One sandwich for breakfast and one sandwich for lunch.

INTERVENTIONS:
Dietary Supplement: Sandwich with butter-like dairy product (40g milk fat) with intact MFGM. One sandwich for breakfast and one sandwich for lunch. — 1) Sandwich with butter-like dairy product (40g milk fat) with intact MFGM.
  Arms: High-fat meal with intact MFGM
Dietary Supplement: Sandwich with butter-like dairy product (40g milk fat) with disrupted MFGM. One sandwich for breakfast and one sandwich for lunch. — 2) Sandwich with butter-like dairy product (40g milk fat) with disrupted MFGM.
  Arms: High-fat meal with destroyed MFGM
Dietary Supplement: Sandwich with butter-like dairy product (40g milk fat) without MFGM. One sandwich for breakfast and one sandwich for lunch. — 3) Sandwich with butter-like dairy product (40g milk fat) without MFGM.
  Arms: High-fat meal without MFGM

SUMMARY:
The aim of the study is to investigate the effects of milk fat globule membrane (MFGM) content and intactness on postprandial metabolic response to a high-fat meal in humans.

The investigators hypothesize that MFGM content and intactness alters the postprandial lipid profile and substrate metabolism in healthy individuals after consumption of a high-fat meal.

DETAILED DESCRIPTION:
The subjects will be invited for four visits in total: one screening visit and three test days separated by a one-week washout period. At the test days, subjects will consume two high-fat meals composed of milk fat with intact MFGM, destroyed MFGM, and without MFGM, respectively. The first meal will be consumed as breakfast and the second meal will be consumed as lunch. Test meals will be isocaloric and with similar macronutrient composition. The meal will consist of a sandwich with a butter-like dairy product.

The three trial days will be completely alike, besides the interventions.

Subjects will arrive at the research lab the night before test day and stay inside a metabolic chamber to acclimatize.

The participants will have one intravenous (iv.) access placed in the elbow on the three trial days where blood samples will be collected at 15, 30, 60, 90, 120, 150 and 180 min after each test meal (breakfast and lunch).

Immediately after consuming each of the two test meals, the subjects will take 1,500mg paracetamol to determine ventricular emptying rate using the acetaminophen test. After this, the subjects can lay in the bed and watch TV, iPad, or work on their laptop.

Before and every hour after consumption of the test meals, the subjects will be asked to fill out an appetite questionnaire (visual analogue scale). At the end of the day the participants will be offered an "ad libitum meal" to measure if MFGM content and intactness influences ad libitum intake of calories at the next meal.

An one-way mixed model of linear regression will be used to compare postprandial area under the curve, ventricular emptying, and ad libitum food intake between the three test days. Secondary outcomes will be analyzed using a two-way mixed model of linear regression with repeated measurements.

Based on the results from a previous study that investigated the effects of the fat and protein structure in dairy products on postprandial triglycerides (20), the investigators will need 11 subjects to detect a 15% decrease in postprandial triglyceride AUC (α=0.05, β=0.80). To account for potential missing values, 12 subjects will be included in total.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Written and informed consent
* HbA1c < 48 mmol/l

Exclusion Criteria:

* Medicine with an impact on blood glucose, lipid profile, or blood pressure and birth control pills
* BMI > 30kg/m2
* Affected screening blood sample as evaluated by the clinical responsible investigator
* Severe claustrophobia
* Lactose intolerance
* Doesn't speak and understand Danish
* Commitment to special diets

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Difference in postprandial triglycerides measured as area under the curve (AUC). | -60 to 180 minutes after first intervention (first meal), 0-180 minuter after second intervention (second high-fat meal)
  Difference in triglycerides AUC after the intervention between high-fat meal with intact MFGM, high-fat meal with destroyed MFGM, and high-fat meal without MFGM.

SECONDARY OUTCOMES:
Difference in concentration of GLP-1 | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of Ghrelin | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of LEAP2 | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of FFA | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of Insulin | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of glucagon | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of cholesterol (total, LDL and HDL) | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of GIP | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of CCK | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration concentration of Gastrin | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration concentration of GDF15 | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of LPS-BP (Lipopolysaccharide Binding Protein) | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration concentration of Cytokines | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of apoB48 | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in concentration of apoB100 | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
Difference in glucose concentration | -60 to 360 minutes after first intervention (first high-fat meal)
  Continuous glucose monitoring (CGM)
Difference in appetite sensation | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
  Visual analogue scale (VAS)
Difference in gastric emptying rate | -60 to 180 minutes after first intervention (first high-fat meal), 0-180 minutes after second intervention (second high-fat meal)
  Acetaminophen test
Ad libitum meal test | 420 minutes after start of test day.
  Amount of food (in grams) intake at the end of the test day to measure if MFGM content and intactness influences ad libitum intake of calories at the next meal.
Metabolic rate | 0-420 minutes
  Indirect calorimetry
Substrate metabolism | 0-420 minutes
  Indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Esben Søndergaard, MD, PhD, Study Director — Steno Diabetes Center Aarhus, Denmark
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No